CLINICAL TRIAL: NCT03505450
Title: Effects of Population Compared to Purposive Sampling for Consensus in an Online Delphi Study
Status: Completed | Type: Observational
Sponsor: ThinkWell (Other)
Responsible Party: Sponsor
Other Study IDs: PLOT-D Sampling Type Effects
Record Dates: First submitted 2018-04-01; First posted 2018-04-23 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Behavior, Consumer
Keywords: decision support tools,
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population sample
  Interventions: Other: Population Sample
- Purposive Sample
  Interventions: Other: Purposive sample

INTERVENTIONS:
Other: Population Sample — full sample of recruited participants
  Groups: Population sample
Other: Purposive sample — purposive sample of recruited participants
  Groups: Purposive Sample

SUMMARY:
This study will be nested as a randomized controlled trial within an online Delphi and will assess the effects of the population sampling compared to purposive sampling for consensus in an online Delphi.

DETAILED DESCRIPTION:
The Delphi method of engaging panels of experts from specific interest areas has been widely utilized in the for the development of research reporting guidelines, core outcome sets, clinical medicine, nursing practice, medical education and healthcare services. An assessment completed by Atkins and colleagues in 2005 report that a small panel of similarly trained experts can develop reliable criteria that inform judgment and support effective decision-making. Despite the wide applicability of the Delphi methodology, it is not known how the number of participants or their similarity as a stakeholder group influences results in an online Delphi.Purposeful sampling will be used with a randomized sample taken from each stakeholder group for analysis and this analysis will be presented alongside the full analysis and the results compared.

The Protocol Lab for Online Trials-Delphi (PLOT-D), which will use an online 3-round Delphi combined with participatory action research to inform the development of a multi-use protocol template for writing protocols for self-recruited online trials of interventional self-management. The Protocol lab will use the Delphi findings, along with earlier research to redesign a series of protocols for online randomized trials with the aim of providing support for citizens to work alongside researchers to build participatory health trials online.

ELIGIBILITY:
Inclusion Criteria:

* Protocol lab online trials Delphi (PLOT-D) Participant

Exclusion Criteria:

* None if meets inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults from an online cohort who are invited to come to consensus in an online Delphi
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Delphi response rate differences as measured by % of completed questions between samples | Up to 20 weeks or study completion
  Full Delphi sample compared to a 10% randomized stratified sample taken from of the 5 stakeholder groups

CONTACTS AND LOCATIONS:
Overall Officials: Amy Price, PhD, Principal Investigator — University of Oxford
Locations (1):
- ThinkWell, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Aggregated data available by request from the study investigator
Supporting Information: Study Protocol, ICF
Time Frame: Post-publication for 5 years
Access Criteria: Contact study investigator by email

REFERENCES:
- [Background] Brookes ST, Chalmers KA, Avery KNL, Coulman K, Blazeby JM; ROMIO study group. Impact of question order on prioritisation of outcomes in the development of a core outcome set: a randomised controlled trial. Trials. 2018 Jan 25;19(1):66. doi: 10.1186/s13063-017-2405-6. PMID 29370827
- [Background] Sinha IP, Smyth RL, Williamson PR. Using the Delphi technique to determine which outcomes to measure in clinical trials: recommendations for the future based on a systematic review of existing studies. PLoS Med. 2011 Jan 25;8(1):e1000393. doi: 10.1371/journal.pmed.1000393. PMID 21283604
- [Background] Fletcher AJ, Marchildon GP. Using the Delphi Method for Qualitative, Participatory Action Research in Health Leadership. International Journal of Qualitative Methods 2014;13:1-18
- [Background] Brice A, Price A, Burls A. Creating a database of internet-based clinical trials to support a public-led research programme: A descriptive analysis. Digit Health. 2015 Nov 20;1:2055207615617854. doi: 10.1177/2055207615617854. eCollection 2015 Jan-Dec. PMID 29942546
- [Background] Bagley HJ, Short H, Harman NL, Hickey HR, Gamble CL, Woolfall K, Young B, Williamson PR. A patient and public involvement (PPI) toolkit for meaningful and flexible involvement in clinical trials - a work in progress. Res Involv Engagem. 2016 Apr 27;2:15. doi: 10.1186/s40900-016-0029-8. eCollection 2016. PMID 29062516
- [Background] Price A, Albarqouni L, Kirkpatrick J, Clarke M, Liew SM, Roberts N, Burls A. Patient and public involvement in the design of clinical trials: An overview of systematic reviews. J Eval Clin Pract. 2018 Feb;24(1):240-253. doi: 10.1111/jep.12805. Epub 2017 Oct 27. PMID 29076631